CLINICAL TRIAL: NCT04149899
Title: A Phase 1/2a Assessment of WB007 Ophthalmic Solution in Subjects With Primary Open-Angle Glaucoma or Ocular Hypertension
Brief Title: Safety and IOP-Lowering Effects of WB007
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: WB007-001
Record Dates: First submitted 2019-10-30; First posted 2019-11-04 (Actual); Results first posted 2023-03-24 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Glaucoma, Primary Open Angle; Ocular Hypertension
Keywords: POAG; OHT; Primary open-angle glaucoma; ocular hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension

STUDY DESIGN:
Intervention Model Description: Part 1 - Open-labelled, single dose, 3-period dose escalation; Part 2 - Double-masked, randomized, parallel comparison
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Part 1 - not masked; Part 2 - Double-masked - neither investigator, study staff nor study participant were aware of treatment assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Part 1 (Period 1): WB007 0.05% (Experimental): WB007 0.05%, single dose to study eye on Day 1
  Interventions: Drug: WB007 0.05%
- Part 1 (Period 2): WB007 0.15% (Experimental): WB007 0.15%, single dose to study eye on Day 1
  Interventions: Drug: WB007 0.15%
- Part 1 (Period 3): WB007 0.4% (Experimental): WB007 0.4%, single dose to study eye on Day 1
  Interventions: Drug: WB007 0.4%
- Part 2: WB007 0.15% (Experimental): WB007 0.15%, dosed twice daily for 14 days
  Interventions: Drug: WB007 0.15%
- Part 2: WB007 0.4% (Experimental): WB007 0.4%, dosed twice daily for 14 days
  Interventions: Drug: WB007 0.4%
- Part 2: Timolol 0.5% (Active Comparator): Timolol 0.5%, dosed twice daily for 14 days.
  Interventions: Drug: Timolol 0.5%

INTERVENTIONS:
Drug: WB007 0.05% — WB007 Ophthalmic Solution 0.05%
  Arms: Part 1 (Period 1): WB007 0.05%
Drug: WB007 0.15% — WB007 Ophthalmic Solution 0.15%
  Arms: Part 1 (Period 2): WB007 0.15%; Part 2: WB007 0.15%
Drug: WB007 0.4% — WB007 Ophthalmic Solution 0.4%
  Arms: Part 1 (Period 3): WB007 0.4%; Part 2: WB007 0.4%
Drug: Timolol 0.5% — Timolol Maleate 0.5% Ophthalmic Solution
  Arms: Part 2: Timolol 0.5%

SUMMARY:
The study evaluated the safety and IOP-lowering effects of WB007 in adults with primary open-angle glaucoma or ocular hypertension in both eyes. This was a 2-part study. Part 1 was a 3-period dose escalation that evaluated 3 concentrations of WB007 ophthalmic solution following a single dose in one eye. Part 2 was a randomized, double-masked, parallel comparison that evaluated two concentrations of WB007 (selected based on Part 1 results) in both eyes compared with timolol 0.5% for 14 days.

ELIGIBILITY:
Inclusion Criteria:

* Ocular hypertension or primary open-angle glaucoma in each eye

Exclusion Criteria:

* History of orthostatic hypotension
* Any active ocular disease
* Anticipated wearing of contact lenses during study
* Contraindication to pupil dilatation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2019-11-14 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2022-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Wirta, MD, Principal Investigator — Eye Research Foundation
Locations (1):
- Eye Research Foundation, Newport Beach, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a 2-part study:
  Part 1: 18 subjects were enrolled and completed study. Based on results from Part 1, two WB007 doses were selected for Part 2.
  Part 2: 59 subjects were enrolled and completed the study.
  No subjects discontinued the study.
Period: Overall Study
Arm/Group | Part 1 (Period 1): WB007 0.05% | Part 1 (Period 2): WB007 0.15% | Part 1 (Period 3): WB007 0.4% | Part 2: WB007 0.15% | Part 2: WB007 0.4% | Part 2: Timolol 0.5%
Started | 6 | 6 | 6 | 23 | 24 | 12
Completed | 6 | 6 | 6 | 23 | 24 | 12
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Part 2: WB007 0.15%: WB007 0.15% dosed twice daily for 14 days
- Part 2: WB007 0.4%: WB007 0.4% dosed twice daily for 14 days
- Total: Total of all reporting groups
Arm/Group | Part 1 (Period 1): WB007 0.05% | Part 1 (Period 2): WB007 0.15% | Part 1 (Period 3): WB007 0.4% | Part 2: WB007 0.15% | Part 2: WB007 0.4% | Part 2: Timolol 0.5% | Total
Number analyzed (Participants) | 6 | 6 | 6 | 23 | 24 | 12 | 77
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.5 (12.44) | 71.2 (4.79) | 77.5 (4.85) | 69.5 (12.88) | 69.0 (13.40) | 64.8 (13.37) | 68.8 (12.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 2 | 14 | 15 | 7 | 46
  Male | 2 | 2 | 4 | 9 | 9 | 5 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 6 | 7 | 1 | 15
  Not Hispanic or Latino | 5 | 6 | 6 | 17 | 17 | 11 | 62
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 6 | 23 | 24 | 12 | 77

OUTCOME MEASURES:

1. Primary Outcome: Part 2: Mean Change From Baseline in Intraocular Pressure (IOP) at Day 14 - Study Eye
Description: IOP is a measurement of the pressure inside the eye and was measured using Goldmann applanation tonometry. Study participants used the study medications in both eyes for 14 days. One eye was designated as the Study Eye at baseline: eyes that met inclusion and exclusion criteria. If both eyes were eligible, the study eye was the eye with higher IOP at Baseline at Hour 0. If both eyes had the same IOP at this timepoint, the right eye was designated as the study eye. IOP was measured at Baseline and Day 14 at Hours 0, 2, 4 and 8. The primary endpoint was the mean change from baseline IOP at Day 14, Hour 2, the timepoint of the peak effect of timolol.
Time Frame: Baseline, Day 14
Population: Modified Intent-to-Treat Population (mITT) with Last Observation Carried Forward: the mITT population consisted of all randomized and treated subjects who provided IOP data at baseline and had at least one post-baseline IOP assessment.
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mm Hg)
Arm/Group | Part 2: WB007 0.15% | Part 2: WB007 0.4% | Part 2: Timolol 0.5%
Number analyzed (Participants) | 23 | 24 | 12
millimeters of mercury (mm Hg)
  Baseline Hour 0 | 26.3 (2.13) | 26.1 (2.17) | 27.1 (3.53)
  Baseline Hour 2 | 24.8 (2.59) | 24.8 (2.16) | 26.7 (4.29)
  Baseline Hour 4 | 25.0 (2.66) | 24.8 (2.27) | 25.8 (4.50)
  Baseline Hour 8 | 24.3 (2.60) | 23.9 (2.00) | 26.1 (4.85)
  Day 14 Hour 0 | -2.6 (2.56) | -3.3 (2.55) | -5.3 (2.93)
  Day 14 Hour 2 | -4.9 (1.85) | -5.1 (2.51) | -6.0 (3.05)
  Day 14 Hour 4 | -4.3 (1.98) | -3.6 (2.94) | -4.0 (3.41)
  Day 14 Hour 8 | -1.8 (2.08) | -1.8 (2.88) | -5.5 (3.33)
Statistical Analysis 1: Comparison: Part 2: WB007 0.15%; A within-group comparison was performed between Baseline, Hour 2 and Day 14, Hour 2, the timepoint for the peak effect of Timolol 0.5%; Test type: Other — The null hypothesis is that the mean change from Baseline, Hour 2 = 0 at Day 14, Hour 2; p < 0.001, t-test, 2 sided — The p-value was not adjusted for multiple comparisons; Mean Difference (Net) = -4.9, 95% CI 2-sided [-5.73 to -4.14], Standard Deviation 1.85
Statistical Analysis 2: Comparison: Part 2: WB007 0.4%; [analysis description as in outcome 1, analysis 1]; Test type: Other — The null hypothesis is that the mean change from Baseline, Hour 2 = 0 at Day 14, Hour 2; p < 0.001, t-test, 2 sided — The p-value was not adjusted for multiple comparisons; Mean Difference (Net) = -5.1, 95% CI 2-sided [-6.14 to -4.02], Standard Deviation 2.51
Statistical Analysis 3: Comparison: Part 2: Timolol 0.5%; [analysis description as in outcome 1, analysis 1]; Test type: Other — The null hypothesis is that the mean change from Baseline, Hour 2 = 0 at Day 14, Hour 2; p < 0.001, t-test, 2 sided — The p-value was not adjusted for multiple comparisons; Mean Difference (Net) = -6.0, 95% CI 2-sided [-7.93 to -4.07], Standard Deviation 3.05
Statistical Analysis 4: Comparison: Part 2: WB007 0.15% vs Part 2: Timolol 0.5%; The mean IOP change from Baseline, Hour 2 to Day 14, Hour 2 (the timepoint for the peak effect of Timolol 0.5%) was compared between WB007 0.15% and Timolol 0.5%; Test type: Non-Inferiority — A pairwise treatment group comparison was performed versus timolol ophthalmic solution 0.5%. A 2-sided 95% confidence interval (CI) for the treatment difference (WB007 minus Timolol) was constructed based on an ANCOVA model. If WB007 was determined to be non-inferior to Timolol, an attempt to show superiority of WB007 over Timolol was made; p = 0.828, ANCOVA — The p-value (2-sided) for superiority was not adjusted for multiple comparisons; The ANCOVA model used the Baseline IOP values at Hour 2 as the covariate; Mean Difference (Net) = 0.14, 95% CI 2-sided [-1.16 to 1.43] — The estimated treatment difference is based on the least-square means from the ANCOVA model
Statistical Analysis 5: Comparison: Part 2: WB007 0.4% vs Part 2: Timolol 0.5%; The mean IOP change from Baseline, Hour 2 to Day 14, Hour 2 (the timepoint for the peak effect of Timolol 0.5%) was compared between WB007 0.4% and Timolol 0.5%; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 4]; p = 0.520, ANCOVA — The p-value (2-sided) for superiority was not adjusted for multiple comparisons; The ANCOVA model used the Baseline IOP values at Hour 2 as the covariate; Mean Difference (Net) = -0.42, 95% CI 2-sided [-1.73 to 0.89] — The estimated treatment difference is based on the least-square means from the ANCOVA model

2. Secondary Outcome: Part 2: Mean IOP at Day 14 - Study Eye
Description: IOP is a measurement of the pressure inside the eye and was measured using Goldmann applanation tonometry. Study participants used the study medications in both eyes for 14 days. One eye was designated as the Study Eye at baseline: eyes that met inclusion and exclusion criteria. If both eyes were eligible, the study eye was the eye with higher IOP at Baseline at Hour 0. If both eyes had the same IOP at this timepoint, the right eye was designated as the study eye. IOP was measured at Baseline and Day 14 at Hours 0, 2, 4 and 8. The primary timepoint was at Day 14, Hour 2, the timepoint of the peak effect of timolol.
Time Frame: Baseline, Day 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mm Hg)
Arm/Group | Part 2: WB007 0.15% | Part 2: WB007 0.4% | Part 2: Timolol 0.5%
Number analyzed (Participants) | 23 | 24 | 12
millimeters of mercury (mm Hg)
  Baseline, Hour 0 | 26.3 (2.13) | 26.1 (2.17) | 27.1 (3.53)
  Baseline, Hour 2 | 24.8 (2.59) | 24.8 (2.16) | 26.7 (4.29)
  Baseline, Hour 4 | 25.0 (2.66) | 24.8 (2.27) | 25.8 (4.50)
  Baseline, Hour 8 | 24.3 (2.60) | 23.9 (2.00) | 26.1 (4.85)
  Day 14, Hour 0 | 23.7 (3.83) | 22.9 (2.42) | 21.8 (1.64)
  Day 14, Hour 2 | 19.9 (2.47) | 19.7 (1.83) | 20.7 (2.18)
  Day 14, Hour 4 | 20.7 (3.10) | 21.2 (2.89) | 21.8 (3.22)
  Day 14, Hour 8 | 22.6 (3.74) | 22.1 (2.52) | 20.6 (3.66)
Statistical Analysis 1: Comparison: Part 2: WB007 0.15% vs Part 2: Timolol 0.5%; The mean IOP for WB007 0.15% was compared to Timolol 0.5% at Day 14, Hour 2, the timepoint for the peak effect of Timolol 0.5% and the primary efficacy timepoint for the study; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 4]; p = 0.828, ANCOVA — The p-value (2-sided) for superiority was not adjusted for multiple comparisons; Mean Difference (Final Values) = 0.14, 95% CI 2-sided [-1.16 to 1.43] — The estimated treatment difference is based on the least-square means from the ANCOVA model
Statistical Analysis 2: Comparison: Part 2: WB007 0.4% vs Part 2: Timolol 0.5%; The mean IOP for WB007 0.4% was compared to Timolol 0.5% at Day 14, Hour 2, the timepoint for the peak effect of Timolol 0.5% and the primary efficacy timepoint for the study; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 4]; p = 0.520, ANCOVA — The p-value (2-sided) for superiority was not adjusted for multiple comparisons; Mean Difference (Final Values) = -0.42, 95% CI 2-sided [-1.73 to 0.89] — The estimated treatment difference is based on the least-square means from the ANCOVA model
Statistical Analysis 3: Comparison: Part 2: WB007 0.15% vs Part 2: Timolol 0.5%; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority — A pairwise treatment group comparison was performed versus timolol ophthalmic solution 0.5%. A 2-sided 95% confidence interval (CI) for the treatment difference (WB007 minus Timolol) was constructed based on an ANOVA model. If WB007 was determined to be non-inferior to Timolol, an attempt to show superiority of WB007 over Timolol was made; p = 0.283, ANOVA — The p-value (2-sided) for superiority was not adjusted for multiple comparisons; The ANOVA model has the treatment group as the main effect; Mean Difference (Final Values) = -0.84, 95% CI 2-sided [-2.39 to 0.71] — The estimated treatment difference is based on the least-square means from the ANOVA model
Statistical Analysis 4: Comparison: Part 2: WB007 0.4% vs Part 2: Timolol 0.5%; [analysis description as in outcome 2, analysis 2]; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 3]; p = 0.189, ANOVA — The p-value (2-sided) for superiority was not adjusted for multiple comparisons; The ANOVA model has the treatment group as the main effect; Mean Difference (Final Values) = -1.02, 95% CI 2-sided [-2.56 to 0.52] — The estimated treatment difference is based on the least-square means from the ANOVA model

ADVERSE EVENTS:
Time Frame: Screening up to Baseline (up to 6 weeks) Part 1: Post-Baseline to Day 2 Part 2: Post-Baseline to Day 14
Description: Adverse Events are reported for all treated subjects.
Arm/Group | Part 1 (Period 1): WB007 0.05% | Part 1 (Period 2): WB007 0.15% | Part 1 (Period 3): WB007 0.4% | Part 2: WB007 0.15% | Part 2: WB007 0.4% | Part 2: Timolol 0.5%
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/23 | 0/24 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/23 | 0/24 | 0/12
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 5/6 | 15/23 | 17/24 | 2/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 (Period 1): WB007 0.05% (N=6) | Part 1 (Period 2): WB007 0.15% (N=6) | Part 1 (Period 3): WB007 0.4% (N=6) | Part 2: WB007 0.15% (N=23) | Part 2: WB007 0.4% (N=24) | Part 2: Timolol 0.5% (N=12)
Instillation Site Pain (General disorders) | 0 | 0 | 0 | 10 | 12 | 1 — General Disorders and Administration Site Conditions
Instillation Site Burn (General disorders) | 0 | 0 | 0 | 2 | 4 | 0 — General Disorders and Administration Site Conditions
Punctate Keratitis (Eye disorders) | 0 | 0 | 5 | 7 | 8 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator shall agree to submit all manuscripts or abstracts to the sponsor for review before submission. Authorship and manuscript composition will reflect joint cooperation between the investigator(s) and sponsor personnel; authorship will be established by mutual agreement, and in line with ICMJE authorship requirements. No individual publications will be allowed prior to completion of the final report of the multicenter study, except as agreed with sponsor.

DOCUMENTS (2):
  • Study Protocol (2021-01-30): https://cdn.clinicaltrials.gov/large-docs/99/NCT04149899/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-02): https://cdn.clinicaltrials.gov/large-docs/99/NCT04149899/SAP_001.pdf